CLINICAL TRIAL: NCT05252065
Title: Cardiac Substructure Radiation Dose and Early Clinical Monitoring of Stage N2-3 Non-Small Cell Lung Cancer Treated With Conventional Radiotherapy
Brief Title: Cardiac Substructure Radiation Dose and Early Clinical Monitoring of Stage N2-3 Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GuizhouMuu
Record Dates: First submitted 2022-01-24; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with NSCLC: all stage N2-3 non-small cell lung cancer patients receive intensity-modulated radiotherapy (IMRT). The prescription dose of PTV is 60-70Gy.
  Interventions: Other: Cardiac biomarkers, Echocardiography,Cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Cardiac biomarkers, Echocardiography,Cardiac magnetic resonance imaging — Troponin I, troponin T, hypersensitive troponin, brain natriuretic peptide and NT-proBNP are detected for cardiac biomarkers;echocardiography and cardiac magnetic resonance imaging are used to measure the functions of heart and vessels.

SUMMARY:
Calculating which cardiac substructure accepting with the highest radiation dose by conventional radiotherapy, then to investigate the relationship between the changes of global longitudinal strain or cardiac magnetic resonance imaging and cardiac biomarkers and the certain cardiac substructure for stage N2-3 non-small cell lung cancer

DETAILED DESCRIPTION:
All patients receive intensity-modulated radiotherapy (IMRT). The prescription dose of PTV is 60-70Gy，Troponin I, troponin T, hypersensitive troponin, brain natriuretic peptide and NT-proBNP are detected before radiotherapy, at the end of radiotherapy (day 15), at the end of radiotherapy and at 1 month after radiotherapy. Echocardiography was performed before radiotherapy, in the middle of radiotherapy (day 15) and at the end of radiotherapy to obtain global longitudinal strain value. Cardiac magnetic resonance imaging is used to measure the blood flow of the anterior descending coronary artery before and at the end of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at TNM stage N2-N3 NSCLC confirmed by histopathology or cytology using IASLC International TNM staging standard (8th edition)
2. KPS score >80; Aged 18 to 75 year-old
3. No contraindications to radiotherapy
4. No history of heart disease before treatment
5. Patients receiving intensity modulated radiation therapy (IMRT)
6. Patients receiving PTV at a prescription dose of 60-70Gy by IMRT
7. Patients receiving radiotherapy alone and concurrent chemoradiotherapy

Exclusion Criteria:

1. Patients with pleural effusion
2. Patients with serious medical illness or infection
3. Patients with acute myocardial infarction within 6 months
4. In patients with NYHA grade 3-4, baseline LVEF before radiotherapy is below 59%
5. Patients with congenital heart diseases, valvular diseases and arrhythmia
6. Patients with pericardial effusion
7. Patients receiving immunotherapy and drug targeted therapy
8. Patients with a history of anthracycline use

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with stage N2-3 non-small cell lung cancerreceive intensity-modulated radiotherapy (IMRT) from Guizhou medical university affiliated cancer hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of Troponin I, troponin T, hypersensitive troponin, brain natriuretic peptide and NT-proBNP | through study completion, an average of 1 year
  These levels are measured with the Siemens ADVIA Centaur XP Immunoassay System, normal ranges of Troponin I, troponin T, hypersensitive troponin, brain natriuretic peptide and NT-proBNP are 0-0.03 ng/mL, 0-0.01 ng/mL, 0-0.04 ng/mL, 0-100 pg/mL, and 0-125pg/mL respectively
Global longitudinal strain value | through study completion, an average of 1 year
  global longitudinal strain value is obtained by offline analysis of 2-dimensional Echocardiography, reduction of more than 15% in left ventricular systole suggests some degree of cardiotoxicity by European Society of Cardiology 2016
The average flow velocity of the anterior descending coronary artery | through study completion, an average of 1 year
  obtained by phase contrast magnetic resonance arteriography of cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lu, Study Chair — Department of thoracic oncology, Affiliated Cancer Hospital of Guizhou Medical University

IPD SHARING:
Plan to Share IPD: No